CLINICAL TRIAL: NCT02362971
Title: External Validity of a Randomized Controlled Trial in Patients With a Femoral Neck Fracture
Brief Title: External Validity of a Randomized Trial in Patients With a Femoral Neck Fracture
Acronym: EXVAL
Status: Active, not recruiting | Type: Observational
Sponsor: Danderyd Hospital (Other)
Responsible Party: Principal Investigator, Olof Skoldenberg, Associate professor, Danderyd Hospital
Other Study IDs: External validity
Record Dates: First submitted 2015-01-26; First posted 2015-02-13 (Estimated); Last update posted 2016-08-30 (Estimated); Status verified 2016-08

CONDITIONS: Femoral Neck Fracture; Hip Fracture
MeSH Terms: conditions — Femoral Neck Fractures; Hip Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Included: Patients included into the randomized controlled trial
- Non-consenters: Patients eligible for participation in the randomized controlled trial but did not give their informed consent and thus excluded in the randomized controlled trial.
- Excluded: Patients, by different reasons excluded from participation in the randomized controlled trial.

SUMMARY:
The aim of this study is to evaluate the external validity of a randomized controlled trial comparing choice of hip arthroplasty for elderly patients (>80 years) with a displaced femoral neck fracture.

The hypotheses are that patient reported hip function, quality of life are better and healthier in those included in the randomized controlled trial than those excluded. The external validity of the randomized controlled trial is acceptable.

A prospective randomized controlled trial is planned and patients with a displaced femoral neck fracture will be included and randomized between either a hemiarthroplasty or total hip arthroplasty. All patients screened will be included in a prospective cohort study for evaluation of the external validity of the randomized controlled trial. The prospective cohort study will consist of 3 different groups.

Patients included in the randomized controlled trial will form group 1. Patients eligible for the randomized controlled trial but did not give their informed consent and therefore excluded, form group 2.

Patients with a femoral neck fracture which by any reason were excluded form group 3.

Primary endpoint is patient-reported hip function (Harris hip score) and pain on the operated extremity evaluated with VAS (Visual Analogue Scale) and patient reported quality of life evaluated with EuroQol (EQ-5D). Secondary outcome measurement are the frequency of the complications, periprosthetic fracture, dislocation, revision surgery due to wound infection (deep and superficial) and loosening of the components. Baseline data, age, sex, comorbidity, cognitive status, weight, height, motor function, complications and reoperations. Follow up is performed 1-2 years after surgery.

Group 1 is followed up in the ongoing randomized controlled trial by visits to the orthopedic department at Danderyd Hospital. Group 2 and 3 are followed up by telephone interview 1-2 year after surgery.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the external validity of a randomized controlled trial comparing choice of hip arthroplasty for elderly patients (>80 years) with a displaced femoral neck fracture.

The hypotheses are:

1. The patient reported hip function and quality of life are better in those included in the randomized controlled trial than those excluded.
2. Patients included in the study are healthier than those excluded.
3. The external validity of the randomized controlled trial is acceptable, defined as the difference between patients that provide and do not provide their informed consent do not reach clinical significance (a mean difference in Harris hip score of 10 points).

All patients above 80 years old with an acute displaced femoral neck fracture at Danderyds hospital AB during 2009-2016 will be screened and asked for participation in a randomized controlled trial. Those who fulfill the criteria for inclusion and give their informed consent are enrolled in the randomized controlled trial. Patients that will not give their informed consent and those which do not fulfill the inclusion criteria are enrolled in a prospective cohort study for evaluation of the external validity.

The prospective cohort study will consist of 3 different groups. Patients included in the randomized controlled trial study will form group 1. Patients eligible for the randomized controlled trial but did not give their informed consent and therefore excluded, form group 2.

Patients with a femoral neck fracture which by any reason were excluded form group 3.

Follow-up is performed 1-2 years after surgery. Inclusion criteria in the randomized controlled trial.

1. Age above 80 years 2. Acute (<36h) displaced femoral neck fracture. 3. Independent walker 4. Abscence of cognitive impairment (Pfeiffer test >7) 5. Did not fulfill any exclusion criteria Exclusion criteria in the randomized controlled trial

1. Patient with osteoarthritis or rheumatoid arthritis in the fractured hip
2. Pathological fracture
3. Non walker
4. Cognitive impairment (Short Portable Mental Questionnaire <7)
5. Contraindication to total hip replacement due to wound, patients with comorbidities, deemed not suitable for a total hip replacement by the anesthesiologist, severe coagulation disorder, and severe drug abuse.
6. Deemed unsuitable for inclusion by other reason.

   1. Primary endpoint is patient-reported hip function (Harris hip score) and pain on the operated extremity evaluated with VAS (Visual Analogue Scale)
   2. Patient reported quality of life evaluated with EQ-5D.

Secondary outcome:

1. Secondary outcome measurement are the frequency of the complications, periprosthetic fracture, dislocation, revision surgery due to wound infection (deep and superficial) and loosening of the components.
2. Baseline data, age, sex, comorbidity, cognitive status, weight, height, motor function and complications and reoperations.

Secondary outcome measurements are obtained in the medical records.

ELIGIBILITY:
Inclusion Criteria randomized controlled trials:

* Age above 80 years
* Acute (<36h) displaced femoral neck fracture.
* Independent walker
* Abscence of cognitive impairment (Short Portable Mental Questionnaire >7points)
* Did not fulfill any exclusion criteria

Exclusion Criteria randomized controlled trial:

* Patient with osteoarthritis or rheumatoid arthritis in the fractured hip
* Pathological fracture
* Non walker
* Cognitive impairment (Short Portable Mental Questionnaire <7points)
* Contraindication to total hip replacement due to wound, patients with comorbidities, deemed not suitable for a total hip replacement by the anesthesiologist, severe coagulation disorder, and severe drug abuse.
* Deemed unsuitable for inclusion by other reason.

Inclusion into prospective cohort study

* Included into the randomized controlled trial.
* Did not give their informed consent for participation in the randomized controlled trial.
* Patients above 80 years of age excluded from participation in the randomized controlled trial due to fulfillment of exclusion criteria or did not fulfill inclusion criteria.

Exclusion into prospective cohort study

* Age below 80 years of age.

Min Age: 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: A femoral neck fracture in the elderly patient is a common cause of suffering and premature death in an aging population. Femoral neck fractures are mainly a fragility (osteoporotic) fracture, predominantly affecting women after menopause. Included in the study are elderly patients (>80 years) with a displaced femoral neck fracture.
Sampling Method: Non-Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2009-09; Primary Completion 2018-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Harris hip score | Up to 2 years
  Hip function as a patient reported outcome measurement

SECONDARY OUTCOMES:
Baseline data (Preoperative baseline data obtained at admission to the hospital) | 1 day
  Age, sex, date of surgery, type of surgical treatment, surgical approach, time, level of competence of the treating surgeon, American Society of Anesthesiologists grade determined by treating anesthesiologist, surgical time, patients weight and length
Mortality | up to 2 years
Complications (Any reason to reoperation) | up to 4 years years
  Any reason to reoperation most commonly prosthetic dislocation, deep infection, periprosthetic dislocation
EQ-5D | up to 2 years
  Health related quality of life, patient reported outcome

CONTACTS AND LOCATIONS:
Overall Officials: Olof G Skoldenberg, MD, PhD, Principal Investigator — Department of clinical sciences at Danderyds hospital, Karolinska Institutet
Locations (1):
- Orthopaedic department, Danderyd Hospital, Stockholm, Stockholm County, Sweden

REFERENCES:
- [Background] Evidence-based health care: a new approach to teaching the practice of health care. Evidence-Based Medicine Working Group. J Dent Educ. 1994 Aug;58(8):648-53. No abstract available. PMID 7930000
- [Background] Petersen MK, Andersen KV, Andersen NT, Soballe K. "To whom do the results of this trial apply?" External validity of a randomized controlled trial involving 130 patients scheduled for primary total hip replacement. Acta Orthop. 2007 Feb;78(1):12-8. doi: 10.1080/17453670610013367. PMID 17453387
- [Background] Pibouleau L, Boutron I, Reeves BC, Nizard R, Ravaud P. Applicability and generalisability of published results of randomised controlled trials and non-randomised studies evaluating four orthopaedic procedures: methodological systematic review. BMJ. 2009 Nov 17;339:b4538. doi: 10.1136/bmj.b4538. PMID 19920015
- [Background] van den Bekerom MP, Hilverdink EF, Sierevelt IN, Reuling EM, Schnater JM, Bonke H, Goslings JC, van Dijk CN, Raaymakers EL. A comparison of hemiarthroplasty with total hip replacement for displaced intracapsular fracture of the femoral neck: a randomised controlled multicentre trial in patients aged 70 years and over. J Bone Joint Surg Br. 2010 Oct;92(10):1422-8. doi: 10.1302/0301-620X.92B10.24899. PMID 20884982
- [Background] Gao H, Liu Z, Xing D, Gong M. Which is the best alternative for displaced femoral neck fractures in the elderly?: A meta-analysis. Clin Orthop Relat Res. 2012 Jun;470(6):1782-91. doi: 10.1007/s11999-012-2250-6. Epub 2012 Jan 26. PMID 22278852
- [Background] Rothwell PM. External validity of randomised controlled trials: "to whom do the results of this trial apply?". Lancet. 2005 Jan 1-7;365(9453):82-93. doi: 10.1016/S0140-6736(04)17670-8. PMID 15639683